CLINICAL TRIAL: NCT00702065
Title: A Multi-center, Multi-regional Observational Study to Test the Responsiveness of the Validated MusiQoL (Multiple Sclerosis International Quality of Life Questionnaire) Instrument to EDSS Status Changes in Any Form of Multiple Sclerosis (MS) in Patients With or Without Treatment
Acronym: MusiQoL
Status: Completed | Type: Observational
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Other Study IDs: 27904
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis Quality of life
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
This is a multi-center, multi-regional observational,24 month study.

Health-related quality of life data from the MusiQoL instrument and SF-36 instrument will be collected at baseline, M6, M12, M18 and M24 in patients with MS. In addition, physical health outcomes such as expanded disability status scores (EDSS) will be collected every 6 months.

DETAILED DESCRIPTION:
This is a multi-center, multi-regional observational,24 month study.

Health-related quality of life data from the MusiQoL instrument and SF-36 instrument will be collected at baseline, M6, M12, M18 and M24 in patients with MS. In addition, physical health outcomes such as expanded disability status scores (EDSS) will be collected every 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has any form of MS (confirmed by McDonald and/or Poser criteria)
2. Patient is 18 years old or more (inclusive, at time of informed consent).
3. Patient has an EDSS score lower than 7.0 (inclusive, at time of informed consent)
4. Patient can be with or without treatment
5. Patient has read, understood, signed and dated informed consent form
6. Patient is able to fill in the questionnaire by him/herself

Exclusion Criteria:

1. CIS Patient (MS not confirmed by Mc Donald and /or Poser criteria)
2. Patient receives or is planned to receive during the course of this study any investigational drug or experimental procedure
3. Patient suffers from dementia in the opinion of the investigator
4. Patient suffers of major medical or psychiatric illness in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 599 (Actual)
Dates: Start 2007-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
MusiQoL (Multiple Sclerosis International Quality of Life Questionnaire) Score | Month 24

CONTACTS AND LOCATIONS:
Locations (30):
- United States (2):
  - Research Site, Phoenix, Arizona
  - Research Site, Las Vegas, Nevada
- Argentina (2):
  - Reseach site, Buenos Aires
  - Research Site, Buenos Aires
- Australia (4):
  - Research Site, Camperdown
  - Research Site, Melbourne
  - Research Site, New Lambton Heights
  - Research Site, Victoria
- Austria (3):
  - Research Site, Graz
  - Research Site, Linz
  - Research Site, Vienna
- France (2):
  - Research Site, Lomme
  - Research Site, Marseille
- Germany (3):
  - Research Site, Bad Wildbad
  - Research Site, Bochum
  - Research Site, München
- Israel (4):
  - Research Site, Afula
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Holon
- Italy (5):
  - Research Site, Brindisi
  - Research Site, Centro Bologna
  - Research Site, Florence
  - Research Site, Modena
  - Research Site, Palermo
- Research Site, Lorenskog, Norway
- Reseach Site, Málaga, Spain
- Research Site, Izmir, Turkey (Türkiye)
- United Kingdom (2):
  - Research Site, Glasgow
  - Research Site, Nottingham

REFERENCES:
- [Result] Auquier P, et al. Responsiveness of the Multiple Sclerosis International Quality of Life(MusiQoL) questionnaire to changes in disability in subjects with multiple sclerosis: 12-month results. Eur J Neurol 2010;17(Suppl 3):486
- [Result] Auquier P, et al. Responsiveness of the Multiple Sclerosis International Quality of Life and Short Form-36 questionnaires to Expanded Disability Status Scale score changes in subjects with multiple sclerosis: 12-month results of an international observational study. 26th Congress of the European Committee for Treatment and Research in Multiple Sclerosis (ECTRIMS): 13-16 October 2010, Gothenburg, Sweden; P650
- [Result] Auquier P, et al. Responsiveness of the Multiple Sclerosis International Quality of Life questionnaire to Expanded Disability Status Scale score changes in subjects with Multiple Sclerosis: Month 12 results from an international observational study. 13th Annual ISPOR Annual European Congress: November 2010, Prague, Czech Republic; P25667
- [Derived] Baumstarck K, Pelletier J, Boucekine M, Auquier P; MusiQoL study group. Predictors of quality of life in patients with relapsing-remitting multiple sclerosis: a 2-year longitudinal study. Rev Neurol (Paris). 2015 Feb;171(2):173-80. doi: 10.1016/j.neurol.2014.09.005. Epub 2015 Jan 2. PMID 25558798
- [Derived] Boucekine M, Loundou A, Baumstarck K, Minaya-Flores P, Pelletier J, Ghattas B, Auquier P. Using the random forest method to detect a response shift in the quality of life of multiple sclerosis patients: a cohort study. BMC Med Res Methodol. 2013 Feb 15;13:20. doi: 10.1186/1471-2288-13-20. PMID 23414459